CLINICAL TRIAL: NCT07254754
Title: LATE-R Trial. A Phase II, Single-Arm, Open-Label, Multicenter Study to Evaluate the Efficacy of Axicabtagene Ciloleucel in Patients With Late Relapse of Diffuse Large B-Cell Lymphoma
Brief Title: Study to Evaluate the Efficacy of Axicabtagene Ciloleucel in Patients With Late Relapse of Diffuse Large B-Cell Lymphoma
Acronym: LATE-R-GEL-23
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español de Linfomas y Transplante Autólogo de Médula Ósea (Other)
Collaborators: Kite, A Gilead Company (Industry); Evidenze Health España (CRO) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LATE-R-GEL-23
Record Dates: First submitted 2025-07-04; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: DIFFUSE LARGE B-CELL LYMPHOMA
Keywords: lymphoma; axicabtagene; geltamo; DIFFUSE LARGE B-CELL LYMPHOMA; DLBCL; RELAPSE
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma; Recurrence | interventions — axicabtagene ciloleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Axicabtagene ciloleucel (Experimental): Treatment consists of a single dose for infusion containing a dispersion for infusion of CAR-positive viable T cells in one infusion bag. The target dose is 2 × 106 CAR-positive viable T cells per kg of body weight (within a range of 1 × 10E6 - 2 × 10E6 cells/kg), with a maximum of 2 × 10E8 CAR-positive viable T cells for patients 100 kg and above.
  Interventions: Drug: Axicabtagene Ciloleucel

INTERVENTIONS:
Drug: Axicabtagene Ciloleucel — Treatment consists of a single dose for infusion containing a dispersion for infusion of CAR-positive viable T cells in one infusion bag. The target dose is 2 × 106 CAR-positive viable T cells per kg of body weight (within a range of 1 × 106 - 2 × 106 cells/kg), with a maximum of 2 × 108 CAR-positive viable T cells for patients 100 kg and above.

SUMMARY:
Single-arm, open-label, multicenter, phase II trial aiming to include approximately 45 patients over 24 months. Patients will receive axicabtagene ciloleucel infusion and will be followed up to 5 years.

The total duration of the study is therefore of 7 years.

DETAILED DESCRIPTION:
Axicabtagene Ciloleucel , an anti-CD19 chimeric antigen receptor (CAR) T-cell therapy, demonstrated a high rate of durable responses with a manageable safety profile, in patients with relapsed or refractory large B-cell lymphoma (LBCL) after two or more previous therapies. Recently, axicabtagene ciloleucel as demonstrated superior efficacy compared to standard of care (SOC) in 2nd line LBCL patients considered eligible for autologous stem-cell transplantation (ASCT) with primary refractory disease or early relapse (ZUMA-7). In this study, after a median follow-up of 24.9 months, the median event-free survival was 8.3 months in the axicabtagene ciloleucel group and 2.0 months in the standard-care group, and the 24-month event-free survival was 41% and 16%, respectively (hazard ratio, [HR] for event or death, 0.40; 95% confidence interval, 0.31 to 0.51; p<0.001). Some response occurred in 83% of the patients in the axicabtagene ciloleucel group and in 50% of those in the SOC group (with a complete response [CR] in 65% and 32% of the patients, respectively). These data led to the approval of axicabtagene ciloleucel by the American and European regulatory agencies, for patients with LBCL refractory to first-line or relapsing within the first year after completion of induction immunochemotherapy.

More recently, the open-label phase 2 ALYCANTE trial assessed the safety and efficacy of axicabtagene ciloleucel as second-line therapy in patients with primary refractory or early relapsed aggressive B-cell lymphoma who were not deemed candidates for ASCT. Treatment with axicabtagene ciloleucel resulted in high response rates (best overall response 92.5%, best CR = 80.0%) and durable remissions (median PFS, 11 months, median overall survival [OS], not reached), with an acceptable safety profile in this population of patients considered unfit for ASCT.

The above-mentioned trials included only patients who were primary refractory or had relapsed within a year of completing first-line treatment. However, no data are available on the efficacy of axicabtagene ciloleucel in second line for patients relapsing more than one year after completion of induction. Although it is generally assumed that the outcome of these patients is better than that of patients showing early failure, still the outcome is not optimal at all, with at least half of the patients dying from the lymphoma in the next months. The current proposal is aimed at studying a possible role of axicabtagene ciloleucel in this subset of cases.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written Informed Consent Form
2. Age > 18 years
3. Patient who understands and speaks one of the country official languages
4. Histologically proven relapsed or refractory aggressive B-cell non-Hodgkin lymphoma (B-NHL) of the following histology at relapse: diffuse large B-cell lymphoma (DLBCL), high-grade B-cell lymphoma (HGBL) and follicular lymphoma Grade 3B per WHO 2016 classification. Indolent B-NHL who transformed into aggressive B-NHL and were previously treated with R-CHOP-like after transformation are eligible. Primary mediastinal B-cell lymphoma are not eligible.
5. Positron-emission tomography (PET)-positive disease
6. Patients must have received adequate first-line therapy including at a minimum:

   * An anti-CD20 monoclonal antibody (rituximab or obinutuzumab), and
   * CHOP or CHOP-like chemotherapy Note: CHOP-like chemotherapy corresponds to ACVBP, EPOCH, or COPADEM. Dose-reduced CHOP (i.e., miniCHOP) is excluded except for dose-reductions of vincristine due to peripheral neuropathy. Patients who have received additional drugs in combination with CHOP or CHOP-like regimen are eligible.
7. Relapsed disease after first line chemo immunotherapy (full dose of R-CHOP or R-CHOP-like regimen), documented by PET-scan and biopsy:

   • Relapsed disease defined as complete remission to first-line therapy followed by biopsy-proven disease relapse after 12 months and up to 5 years from end of first-line therapy.
8. Patients must meet CAR-T-eligible criteria as defined by:

   * Patient deemed eligible for CAR T-cells therapy by the CAR-T physician
   * AND all the following criteria:

     * ECOG performance status of 0, 1 or 2
     * Adequate vascular access for leukapheresis procedure (either peripheral or central venous line)
     * Absolute neutrophil count (ANC) ≥ 1 x 109/L
     * Platelets ≥ 75 x 109/L
     * Absolute lymphocyte count ≥ 0.1 x 109/L
     * Creatinine clearance (CrCl) as estimated by Cockcroft Gault or MDRD ≥ 40 mL/min
     * Serum alanine aminotransferase/aspartate aminotransferase (ALT/AST) ≤ 2.5xULN
     * Total bilirubin <1.5 mg/dL, except in patients with Gilbert's syndrome
     * Cardiac ejection fraction ≥ 45%
     * Baseline oxygen saturation ≥ 92% on room air
9. Females of childbearing potential must have a negative serum or urine pregnancy test (females who have undergone surgical sterilization or who have been postmenopausal for at least 12 months are not considered to be of childbearing potential).

Exclusion Criteria:

1. Patients who received more than one prior line of systemic therapy
2. Early relapsed disease defined as complete remission to first-line therapy followed by biopsy-proven disease relapse before 12 months from end of first-line therapy.
3. Refractory disease defined as:

   * Progressive disease (PD) during first-line therapy
   * Stable disease (SD) as best response after at least 4 cycles of first-line therapy (e.g., 4 cycles of R-CHOP)
   * Partial response (PR) as best response after at least 6 cycles, and biopsy-proven residual disease
4. Patients who received first line of R-CHOP or obinutuzumab-CHOP for an indolent B-NHL who relapse as transformed aggressive B-NHL after a year from the end of first-line therapy are NOT eligible.
5. Prior CD19 targeted therapy
6. Patients with cardiac atrial or cardiac ventricular lymphoma involvement
7. Requirement for urgent therapy due to tumor mass effects, such as bowel obstruction or blood vessel compression
8. Patient with clinically significant pleural effusion
9. History of another primary malignancy that has not been in remission for at least 3 years (except for nonmelanoma skin cancer or carcinoma in situ (eg, cervix, bladder, breast)). A maintenance treatment is not allowed.
10. Patients with detectable Central Nervous System (CNS) lymphoma. Patients with a history of CNS lymphoma but no active CNS disease (after systematic MRI and lumbar puncture) at the time of enrolment will be eligible.
11. Presence of CNS disorder such as dementia, autoimmune disease with CNS involvement, cerebral edema with confirmed structural defects by appropriate imaging, or seizure disorders requiring active anticonvulsive medication. History of stroke, transient ischemic attack, or posterior reversible encephalopathy syndrome (PRES) within 12 months prior to enrolment.
12. Presence of any indwelling line or drain (eg, percutaneous nephrostomy tube, indwelling Foley catheter, biliary drain, or pleural/peritoneal/pericardial catheter). Ommaya reservoirs and dedicated central venous access catheters, such as a Port-a-Cath or Hickman catheter, are permitted.
13. History of acute or chronic active hepatitis B or C infection (seropositivity). If there is a positive history of treated hepatitis B or hepatitis C (negative HBsAg and positive Anti-HBc/ positive anti-HCV), the viral load HBV DNA/ HCV RNA) must be undetectable per quantitative polymerase chain reaction (PCR) and/or nucleic acid testing
14. Positive for human immunodeficiency virus (HIV) unless taking appropriate anti-HIV medications, with an undetectable viral load by PCR and with a CD4 count > 200 cells/uL.
15. Uncontrolled systemic fungal, bacterial, viral or other infection despite appropriate antimicrobials or other treatment at the time of leukapheresis or axicabtagene ciloleucel administration
16. History of any one of the following cardiovascular conditions within the past 12 months: Class III or IV heart failure as defined by the New York Heart Association, cardiac angioplasty or stenting, myocardial infarction, unstable angina, or other clinically significant cardiac disease
17. Presence of primary immunodeficiency
18. History of any medical condition including but not limited to autoimmune disease (e.g., Crohn's disease, rheumatoid arthritis, systemic lupus) requiring systemic immunosuppression and/or systemic disease modifying agents within the last year. Endocrine conditions that require maintenance with physiologic dose steroids are allowed.
19. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis per chest computed tomography (CT) scan at screening. History of radiation pneumonitis in the radiation field (fibrosis) is allowed.
20. History of severe immediate hypersensitivity reaction to tocilizumab or any of the agents used in this study
21. History of severe, immediate hypersensitivity reaction attributed to aminoglycosides, cyclophosphamide or fludarabine
22. Treatment with a live, attenuated vaccine within 6 weeks prior to initiation of study treatment or anticipation of need for such a vaccine during the study
23. Women of childbearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of lymphodepletion chemotherapy on the fetus or infant.
24. Patients of either sex who are not willing to practice birth control from the time of consent during treatment and for at least 12 months after conditioning chemotherapy dosing or axicabtagene ciloleucel dosing, whichever is later
25. In the investigator's judgment, the patient is unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participation
26. Adult person unable to provide informed consent because of intellectual impairment, any serious medical condition, laboratory abnormality or psychiatric illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Response month 3 | Month 3
  The Complete Metabolic Response, defined as negative findings on a PET/CT scan at month 3 after receiving axicabtagene ciloleucel infusion at day 0. The negativity of PET/CT findings will be assessed according to Lugano Classification and Deauville criteria

SECONDARY OUTCOMES:
Response month 3 central | Month 3
  The Complete Metabolic Response defined as negative findings on a PET/CT scan at month3 after receving axicabtagene ciloleucel infusion as assessed by central imaging review of PET/CT
Overall response rate | Month 3
  The Overall response rate (ORR) defined as the percentage of patients who achieved partial metabolic response (PMR) or complete metabolic response (CMR) according to the Lugano Classification criteria at month 3 determined by both central and investigator assessments.
Best objective response | 1 year
  Best objective response rate defined as the percentage of CMR + PMR determined by the investigator assessment among all patients between month 1 and month 12 from axicabtagene ciloleucel infusion
Best complete response rate | 1 year
  Best Complete Response rate defined as the percentage of CMR determined by the investigator assessment among all patients between month 1 and month 12 from axicabtagene ciloleucel infusion
Overall survival | Up to 5 years
  The overall survival, defined as the time from inclusion to death from any cause. Alive patients will be censored at their last follow-up date.
Progression free survival | Up to 5 years
  The Progresison Free Survival, defined as the time from axicabtagene ciloleucel infusion to the first observation of documented disease progression/relapse (based on investigator disease assessment (INV)) or death due to any cause. If a patient has not progressed or died, PFS will be censored at the time of last visit with adequate assessment
Event Free Survival | Up to 5 years
  Event-free survival (EFS), defined as the time between leukapheresis and to any event preventing axicabtagene ciloleucel infusion if axicabtagene ciloleucel is never infused, or death, disease progression, or instauration of a new lymphoma therapy for lymphoma progression after axicabtagene ciloleucel infusion. Patients without documented event at the time of analysis will be censored at the time of last visit with adequate assessment.
Duration of Response | Up to 5 years
  The Duration of Response (DOR), defined as the time from attainment of PMR or CMR to the date of first documented disease progression/relapse (based on investigator disease assessment) or death from any cause
Duration of Complete Response | Up to 5 years
  Duration of complete response (DoCR), defined as the time from achievement CMR to the date of first documented disease progression/relapse (based on investigator disease assessment) or death from any cause.
Adverse events | Up to 4 weeks
  Type, frequency and severity of adverse events (AEs) and serious adverse events (SAEs)
AESIs | Up to 5 years
  Incidence, severity and treatment of adverse events of special interest: Cytokine release syndrome (CRS), immune effector cell-associated neurotoxicity syndrome (ICANS), prolonged cytopenia and infections, hypogammaglobulinemia and emergent secondary malignancies.
Quality of Life assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) | Up yo 1 year
  The EORTC QLQ-C30 is a 30-item questionnaire measuring cancer patients' physical, emotional, and social functioning. Scores range from 0 to 100. Range: 0 (worst) to 100 (best). Higher scores indicate better quality of life for functional scales and worse symptoms for symptom scales.
Quality of Life assessed using the EuroQol 5-Dimension 5-Level Questionnaire (EQ-5D-5L) | Up to 1 year
  The EQ-5D-5L evaluates mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. It includes a visual analog scale (VAS) from 0 to 100. Range: 0 (worst imaginable health) to 100 (best imaginable health). Higher scores indicate better health status.
Quality of Life assessed using the EORTC Quality of Life Questionnaire for High-Grade Non-Hodgkin Lymphoma (QLQ-NHL-HG29) | Up to 1 year
  The QLQ-NHL-HG29 is a disease-specific module assessing symptoms and functioning in patients with high-grade non-Hodgkin lymphoma. Scores range from 0 to 100. Range: 0 to 100. Higher scores indicate worse symptoms or problems.

OTHER OUTCOMES:
Total Metabolic Tumor | Up to 2 years
  Correlation between Total Metabolic Tumor Volume (TMTV) pre-axicabtagene ciloleucel infusion and efficacy/toxicity
Phenotypic expression of lineage and checkpoint markers in tumor | Up to 2 years
  Histologic, phenotypic, genomic, transcriptomic, and molecular characteristics of Expression of CD19, CD20, CD79a, PD-L1 and other protocol-specified markers assessed by IHC or immunofluorescence on tumor tissue pre- and post-treatment.
Cytokine levels | Up to week 4
  Concentrations of predefined cytokines (e.g., IL-6, IFN-γ, TNF-α) measured in serum pre-treatment and at specified post-treatment time points.Unit of Measure: Picograms per milliliter (pg/mL).
Minimal residual disease | Up to 2 years
  Minimal residual disease assessment by ctDNA
Immune-escape mechanisms | Up to 2 years
  Immune-escape mechanisms including resistance of tumor cells to T-cell killing and tumor-induced immune suppression
Immune cell subset frequencies in blood | Up to 2 years
  Relative frequencies of immune cell subsets (e.g., CD3+ T cells, CD4+, CD8+, regulatory T cells, NK cells) by flow cytometry at scheduled times.Unit of Measure: Percentage of peripheral blood mononuclear cells (% of PBMC) or cells per microliter (cells/µL).

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Bastos-Oreiro, Principal Investigator — Hospital General Universitario Gregorio Marañón; Alejandro Martín García-Sancho, Principal Investigator — Hospital Universitario Salamanca; Armando López-Guillermo, Principal Investigator — Hospital Clinic of Barcelona
Locations (15):
- Spain (15):
  - Complejo Hospitalario Universitario A Coruña, A Coruña, A Coruña
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario de Salamanca, Salamanca, Castille and León
  - Hospital Universitari Vall d'Hebron, Barcelona, Catalonia
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Catalonia
  - Institut Català d'oncologia de L'Hospitalet, L'Hospitalet de Llobregat, Catalonia
  - Hospital Universitario Donostia, San Sebastián, Gipuzkoa
  - Complejo Hospitalario Universitario de Gran Canaria Dr. Negrín, Las Palmas de Gran Canaria, Las Palmas
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital General Universitario Morales Meseguer, Murcia, Murcia
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario Virgen del Rocío, Seville, Sevilla
  - Hospital Clínico Universitario de Valencia, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in hematology diseases.
  All individual data collected during the trial will be available. Data shared will be coded, with no PHI included. Study protocol, statistical analysis plan, informed consent form and clinical study report will be also available. Information will be available beginning 6 months after final publication with no end date established. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party. Data requests can be submitted starting 6 months after article publication. Access to trial IPD can be requested by qualified researchers and will be provided following review and approval of a research and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact to GELTAMO though the web page: https://www.geltamo.com/contacto

REFERENCES:
- See also: GELTAMO web page — https://www.geltamo.com/